CLINICAL TRIAL: NCT06666959
Title: Comparison of the Neuroprotective Effect of Sevoflurane Versus Propofol in Patients Undergoing Endovascular Coiling of Cerebral Aneurysm
Brief Title: Sevoflurane Versus Propofol in Endovascular Coiling of Cerebral Aneurysm
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, mingxin zhu, associate professor, Tongji Hospital
Other Study IDs: TJ-IRB20230413; SW-001 (Other: department of neurosurgery in Tongji hospital)
Record Dates: First submitted 2024-10-26; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Propofol; Sevoflurane
MeSH Terms: interventions — Anesthetics; Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- patients undergoing endovascular coiling of cerebral aneurysm in Tongji hospital: The present clinical study was carried out with the aim of determine whether the inflammatory effect differs when using propofol or sevoflurane anesthesia.
  Interventions: Drug: Anesthesia Agent

INTERVENTIONS:
Drug: Anesthesia Agent — intravenous anesthetic and inhalation anesthetic
  Other Names: sevoflurane; propofol

SUMMARY:
The goal of this observational study is to learn about the anti-inflammatory effects of anesthetics on patients undergoing endovascular coiling of cerebral aneurysm. The main question it aims to answer is:

Does sevoflurane or propofol affect the inflammatory response in subarachnoid hemorrhage?

Participants already undergoing endovascular coiling of cerebral aneurysm will have their serum levels of inflammatory factors measured.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18 years and older presenting to the Tongji hospital for endovascular coiling of cerebral aneurysm were eligible for enrollment.

Exclusion Criteria:

* have an endocrine system disease
* pregnancy
* have other brain disorders
* take drugs that alter endocrine hormones
* receive perioperative blood derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Tongji hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Concentration of interleukin-10 | From enrollment to 3 months postoperation
  Test the concentration of interleukin-10 of the participants

SECONDARY OUTCOMES:
Concentration of interleukin-1 | From enrollment to 3 months postoperation
  Test the Concentration of interleukin-1 in participants
Concentration of interleukin-2 | From enrollment to 3 months postoperation
  Test the concentration of interleukin-2 in participants
Concentration of interleukin-6 | From enrollment to 3 months postoperation
  Test the concentration of interleukin-6 in participants
Concentration of interleukin-8 | From enrollment to 3 months postoperation
  Test the concentration of interleukin-8 in participants
Concentration of tumor necrosis factor | From enrollment to 3 months postoperation
  Test the concentration of tumor necrosis factor in participants
Concentration of S100B | From enrollment to 3 months postoperation
  Test the concentration of S100B in participants
length of stay | through study completion, an average of 6 months
  The time from admission to discharge
costs | through study completion, an average of 6 months
  Hospitalization expenses
Glasgow Coma Score | From enrollment to 3 months postoperation
  The scores are ranging from 3 to 15. And higher scores mean a betterr outcome .

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Wuhan, Hubei, China